CLINICAL TRIAL: NCT01994642
Title: A Randomized, Double-Blind, Parallel Design, Multiple-Site Study to Evaluate the Clinical Equivalence of Ciprofloxacin 0.3%/Dexamethasone 0.1% Sterile Otic Suspension (Par) Compared to CIPRODEX® (Ciprofloxacin 0.3%/Dexamethasone 0.1%) Sterile Otic Suspension (Alcon) in the Treatment of Acute Bacterial Otitis Media in Children With Patent Tympanostomy Tubes
Brief Title: Bioequivalence of Two Ciprofloxacin 0.3%/Dexamethasone 0.1% Sterile Otic Suspensions in Otitis Media in Children With Tympanostomy Tubes
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: FDA's draft guidance (revised March 2015) provided two options for determining bioequivalence: 1) in-vitro or 2) in-vivo studies
Sponsor: Par Pharmaceutical, Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 71205503
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2017-09-26 (Actual); Status verified 2017-09

CONDITIONS: Otitis Media in Patients With Tympanostomy Tubes
MeSH Terms: interventions — Ciprofloxacin; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Reference (Active Comparator): CIPRODEX® (ciprofloxacin 0.3%/dexamethasone 0.1%)
  Interventions: Drug: CIPRODEX® (ciprofloxacin 0.3%/dexamethasone 0.1%)
- Placebo (Placebo Comparator): Placebo Sterile Otic Suspension
  Interventions: Drug: Placebo Sterile Otic Suspension
- Test (Experimental): Ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension
  Interventions: Drug: Ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension

INTERVENTIONS:
Drug: Ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension
  Arms: Test
Drug: CIPRODEX® (ciprofloxacin 0.3%/dexamethasone 0.1%)
  Arms: Reference
Drug: Placebo Sterile Otic Suspension
  Arms: Placebo

SUMMARY:
The objective of this study is to compare the relative efficacy and safety of the test formulation of ciprofloxacin 0.3%/dexamethasone 0.1% sterile otic suspension (Par) to the already-marketed formulation CIPRODEX® (ciprofloxacin 0.3%/dexamethasone 0.1%) sterile otic suspension (Alcon) in the treatment of acute bacterial otitis media in children with patent tympanostomy tubes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 6 months-12 years of age inclusive.
2. Parent or legal guardian has signed informed consent form, which meets all of the criteria of current FDA regulations.
3. Based on the patient's age, comprehension and communication developmental skills has provided assent to participate in an appropriate format.
4. Confirmed insertion of a patent tympanostomy tube(s) in the infected ear(s).
5. Clinical signs and symptoms consistent with acute bacterial otitis media in at least one ear and a score of at least 2 for otorrhea using the following scale 0=none, 1=mild, 2=moderate, 3=severe, (see Appendix A for rating scale and severity definitions).
6. Otorrhea has been present for 21 days or less.
7. The presence of infection confirmed by a positive bacterial culture for the presence of Staphylococcus aureus, Streptococcus pneumoniae, Haemophilus influenzae, Moraxella catarrhalis or Pseudomonas aeruginosa. As the results of the bacterial culture will not be immediately known, patients who meet all the other inclusion/exclusion criteria may be enrolled in the study pending the results of the bacterial culture.

Exclusion Criteria:

1. Tympanostomy tube placement occurred within 3 days or less of screening visit.
2. Tympanostomy tubes containing silver oxide or silver salts, or T-type tubes.
3. Signs and symptoms of otitis media for longer than 21 days prior to being screened for inclusion in the study.
4. Since the insertion of the tympanostomy tube(s), more than 1 previous episode of otitis media within the previous 3 months or more than 4 episodes within the previous 12 months.
5. Provided any therapeutic drug treatment for current episode of otitis media within the previous 14 days.
6. Current or previous history of any otologic surgery other than insertion/removal of tympanostomy tubes in infected ear(s).
7. Clinical diagnosis that suggests current signs or symptoms are not caused by acute bacterial otitis media e.g. otitis externa
8. Clinical diagnosis of malignant otitis externa
9. Mastoid cavities, stenosis, exostosis or tumors of either ear or other noninfectious diseases of either ear.
10. Suspected concurrent fungal or viral infection (e.g. herpes simplex) of either ear.
11. Dermatitis of the infected ear such as psoriasis or seborrhea that would complicate evaluations.
12. Any known hypersensitivity to ciprofloxacin or other carboxyquinolone derivatives, dexamethasone or corticosteroids or other ingredients of the formulation.
13. Significant underlying disease such as diabetes, HIV or other immunocompromised conditions or receiving therapy that may cause patient to be immunocompromised.
14. Significant history or current evidence of chronic infectious disease, system disorder, organ disorder or other medical condition that in the Investigator's opinion would place the study patient at undue risk by participation or could jeopardize the integrity of the study evaluations.
15. Investigator believes that severity of infection is such that systemic antibiotics would be the preferred treatment option.
16. Use of any systemic antibacterial products or topical antibacterial products in the ear(s) within 14 days of screening for the study.
17. Use of any systemic anti-inflammatory products or topical anti-inflammatory products in the ear(s) (such as corticosteroids and NSAIDs) within 7 days of screening for the study.
18. Use of any topical or otic medication in the affected ear within 7 days prior to screening.
19. Use of any astringents such as vinegar, alcohol or medicated cleansing or swabbing of the ear within 48 hours of the baseline bacterial culture swab.
20. Receipt of any drug or device as part of a research study within 30 days prior to dosing.
21. Previous participation in this study.

Ages: 6 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 203 (Actual)
Dates: Start 2013-11; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Clinical Success | Day 14-21
  A patient who is considered a "clinical success" at Visit 4 (Test of Cure/End of Study) will have no signs or symptoms of active AOMT that were present at baseline nor any new signs or symptoms of AOMT have developed

SECONDARY OUTCOMES:
Cessation of Otorrhea | Day 14-21

CONTACTS AND LOCATIONS:
Overall Officials: Chandra Vattikonda, Ph.D., Study Director — Par Pharamceutical, Inc.
Locations (23):
- United States (23):
  - Birmingham Pediatrics, Birmingham, Alabama
  - Agave Clinical Ressearch, Mesa, Arizona
  - Arizona Center for Clinical Trials, Phoenix, Arizona
  - Visions Clinical Research, Tuscon, Tucson, Arizona
  - Alliance Research, Long Beach, California
  - San Marcus Research Clinic, Miami, Florida
  - Florida Medical Center and Research Inc., Miami, Florida
  - South Miami Clinical Research Group, Miami, Florida
  - Miami Dade Medical Resarch Institute, Miami, Florida
  - Global Health Research Center, Miami Lakes, Florida
  - Winter Park Clinical Research, Winter Park, Florida
  - Research Integrity, Owensboro, Kentucky
  - Dr. Craig Spiegel, Bridgeton, Missouri
  - Dr. Scott Mathei, Henderson, Nevada
  - Piedmont Ear Nose and Throat Associates, PA, Winston-Salem, North Carolina
  - Accecss MD, Clinical Resarch, Huber Heights, Ohio
  - Cyn3gry, Gresham, Oregon
  - Rainbow Research, Inc, Barnwell, South Carolina
  - Dr. John Ansley, Orangeburg, South Carolina
  - Spartanburg and Greer ENT, Spartanburg, South Carolina
  - PMG Research of Bristol, Bristol, Tennessee
  - Eagle Family Medical Associates, Crossville, Tennessee
  - The Education and Research Foundation, Inc, Lynchburg, Virginia